CLINICAL TRIAL: NCT03069924
Title: Gain-framed Messages and NRT Sampling to Promote Smoking Cessation in Lung Cancer Screening Programs
Brief Title: Gain-framed Messages and NRT for Lung Cancer Screening Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Benjamin Toll, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00055397; 5R01CA207229-06 (NIH)
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Results first posted 2024-11-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Lung Cancer Screening; Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Unframed Messaging (Active Comparator): Unframed smoking cessation materials
  Interventions: Combination Product: Unframed messaging materials
- Gain-framed Messaging (Experimental): Gain-framed messaging
  Interventions: Behavioral: Gain-framed messaging

INTERVENTIONS:
Behavioral: Gain-framed messaging — Gain-framed messaging materials
  Arms: Gain-framed Messaging
Combination Product: Unframed messaging materials — Unframed smoking cessation materials
  Arms: Unframed Messaging

SUMMARY:
This research is a randomized smoking cessation trial conducted within and specifically personalized for lung cancer screening patients presenting to a lung screening clinic. Novel tobacco treatments for this population are critically needed, given the growing population of lung screening patients, which will grow dramatically now that lung screening is an approved CMS benefit. In the proposed study, we will test a gain-framed messaging intervention specifically designed for lung screening patients (vs. unframed messaging), as well as evaluating NRT sampling (vs. no medication) at 2 study sites. Our project is designed to be translational (in that it can be transferable from our controlled efficacy study to other lung screening programs).

ELIGIBILITY:
Inclusion Criteria:

1. 50 years or older
2. at least a 20-pack year history of smoking
3. current smoker (defined as any smoking in the past 30 days)
4. willing to be randomized
5. English speaking

Exclusion Criteria:

1. unstable psychiatric/medical conditions such as suicidal ideation, acute psychosis, severe alcohol dependence, or dementia,
2. known allergy to adhesives
3. being in the immediate (within 2 weeks) post myocardial infarction period
4. serious arrhythmias
5. unstable angina pectoris
6. hemodynamically or electrically unstable.
7. current participation in another tobacco treatment program (e.g., using medication from a primary care doctor, Quitline, etc.)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2024-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Toll, PhD, Principal Investigator — Medical University of South Carolina; Alana Rojewski, PhD, Study Director — Medical University of South Carolina
Locations (2):
- United States (2):
  - Yale Cancer Center, New Haven, Connecticut
  - Medical University of South Carolina, Charleston, South Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Gain-framed Messaging: Gain-framed messaging
  Gain-framed messaging : Gain-framed messaging materials
Period: Overall Study
Arm/Group | Unframed Messaging | Gain-framed Messaging
Started | 183 | 184
Completed | 126 | 116
Not Completed | 57 | 68

BASELINE CHARACTERISTICS:
Population: Baseline population consists of all consented and randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Unframed Messaging | Gain-framed Messaging | Total
Number analyzed (Participants) | 183 | 184 | 367
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 127 | 115 | 242
  >=65 years | 56 | 69 | 125
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.2 (5.6) | 62.7 (6.0) | 62.4 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 102 | 210
  Male | 75 | 82 | 157
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 8
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 66 | 56 | 122
  White | 102 | 115 | 217
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 8 | 19
Region of Enrollment [Number; unit: participants]
  United States | 183 | 184 | 367
Cigarettes Smoked Per Day [Mean (Standard Deviation); unit: Cigarettes Smoked Per Day, Average] | 15.6 (7.8) | 15.6 (8.2) | 15.6 (8.0)
Abstinent at Study Baseline [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Smoking Cessation - Available Data
Description: Gain-framed messaging vs. Unframed messaging. 7-day, self-reported abstinence from cigarettes at the 6- month follow-up visit
Time Frame: 6 month follow-up
Population: All available participants are included in the analysis of 7 day point prevalence abstinence at the 6-month follow up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Unframed Messaging | Gain-framed Messaging
Number analyzed (Participants) | 126 | 116
Participants | 15 | 19

2. Secondary Outcome: Cigarettes Smoked Per Day - Average
Description: Gain-framed messaging vs. Unframed messaging - average reported cigarettes smoked per day.
Time Frame: 6 month follow-up
Population: all participants with data available at the 6-month follow up visit.
Measure: Mean (95% Confidence Interval); unit: Average Cigarettes Smoked Per Day
Arm/Group | Unframed Messaging | Gain-framed Messaging
Number analyzed (Participants) | 126 | 116
Average Cigarettes Smoked Per Day | 9.7 [8.3 to 11.1] | 8.9 [7.5 to 10.3]

3. Secondary Outcome: Smoking Cessation - Imputed
Description: Gain-framed messaging vs. Unframed messaging. 7-day, self-reported abstinence from cigarettes at the 6- month follow-up visit. Missing participant data imputed to no cessation. 3 participants from the unframed group were not included as they had died prior to the 6-month visit.
Time Frame: 6 Month Follow up Visit
Population: all randomized participants whom were alive at the 6-month follow up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Unframed Messaging | Gain-framed Messaging
Number analyzed (Participants) | 180 | 184
Participants | 15 | 19

ADVERSE EVENTS:
Time Frame: Adverse events were collected from study entry to the conclusion of the 6-month follow up session or when a participant withdrew from the study.
Arm/Group | Unframed Messaging | Gain-framed Messaging
All-Cause Mortality (participants affected / at risk) | 3/183 | 0/184
Serious Adverse Events (participants affected / at risk) | 0/183 | 0/184
Other Adverse Events (participants affected / at risk) | 0/183 | 0/184

LIMITATIONS AND CAVEATS:
Due to low accrual for this clinical trial during the COVID pandemic, we worked with our study statistician and NCI Program Officer to collapse our 4 arm trial to 2 arms. This allowed us to meet our accrual goal and complete the study while still retaining the ability to test our Primary Aim.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT03069924/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT03069924/ICF_001.pdf